CLINICAL TRIAL: NCT03441763
Title: Impact of Body Weight on Shifting of Foot Pressure Among Obese Subjects
Brief Title: Shifting and Distribution of Foot Pressure Among Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Alsayed Abd Elhameed Shanb, Associate Professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-03-065
Record Dates: First submitted 2017-04-12; First posted 2018-02-22 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Foot pressure, Obese, and normal Subjects
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal participants (Experimental): Emed foot device 3 times/measure to determine foot pressure in normal participants. .
  Interventions: Device: Emed foot device
- Over weight participants (Experimental): Emed foot device 3 times/measure to determine foot pressure in over weight participants.
  Interventions: Device: Emed foot device
- Obese participants (Experimental): Emed foot device 3 times/measure foot pressure in obese participants.
  Interventions: Device: Emed foot device

INTERVENTIONS:
Device: Emed foot device — foot pressure will be measure by using emed foot pressure system

SUMMARY:
Background: The foot is considered a sensitive structure of musculoskeletal system that bears significant loads of the body weight during walking. So, the evaluation of the body weights on planter pressure distribution during walking among adult obese subjects is very critical for foot dysfunctions.The aims:To evaluate the planter pressure distribution in normal ,over weight and obese adult during dynamic situation. Subjects and Methods: A one-hundred fifty normal adult (male and female) subjects will be recruited in this study. They will be divided into Group-I: includes 50 normal subjects Group-II: includes 50 of over weight subjects.group-III 50 obese adult subjects The all three groups will be detected according to the individual BMI. The details of the study will be explained to each participant and a consent form was signed by each subject.Each participant should be free from any musculoskeletal or locomotors disorders Conclusion: Results of this study can help physical therapists to understand the foot pressure distribution map for normal , over weight and obese and non-obese subjects to detect any foot abnormalities and detect any causes of foot dysfunctions.

DETAILED DESCRIPTION:
A one hundred fifty volunteers (male and female), age from 20 to 40 years old subjects will be recruited in this study. Demographic data of all participating subjects like age, weight, height, feet size, and body mass index (BMI) will be assessed. All participants will be assigned to three groups per measurement of individual BMI: Group-I: includes 50 normal subjects (18.5 -24.9 BMI); Group-II: includes50 overweight subjects (25.0 -29.9 BMI); Group-III: includes 50 obese subjects (30.0 and Above BMI) (Nuttall, 2015). The procedure and purpose of the study will be explained in details for all participants. A consent form will be signed by each participant. Human research already approved by Institutional review board of Imam Abdulrahman Bin Faisal University(University of dammam previously ).IRB.2017- 03-065.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are normal or over weight or obese . Subjects who are free from any musculoskeletal abnormalities .

Exclusion Criteria:

Subjects has any foot deformity, flat foot, acute lower extremity trauma, lower extremity surgery like prosthesis operations of the hip, knee, ankle or foot, Subjects has problems of cooperation including; eye, ear oar cognitive disorders, diabetes or related peripheral neuropathy, vascular insufficiency, walking aids .

Subjects has age greater than 40 or less than 25 years.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Foot planter pressure | 3 months
  Foot plantar pressure during walking will be detected in four anatomical foot areas (hindfoot, midfoot, forfoot, toes) for 150 normal and obese person using Emed pressure system

CONTACTS AND LOCATIONS:
Overall Officials: Alsayed A Shanb, PhD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- University of Dammam, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The final results only will be shared

REFERENCES:
- [Background] Stess RM, Jensen SR, Mirmiran R. The role of dynamic plantar pressures in diabetic foot ulcers. Diabetes Care. 1997 May;20(5):855-8. doi: 10.2337/diacare.20.5.855. PMID 9135955
- See also: doi: 10.1016/j.gaitpost.2008.01.012. Epub 2008 M — http://www.ncbi.nlm.nih.gov/pubmed/18337103